CLINICAL TRIAL: NCT01989338
Title: Effects of Hallux Valgus Deformity on Rear Foot Position, Pain, Function, and Quality of Life in Women
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Gursoy Coskun, Hacettepe University, Hacettepe University
Other Study IDs: LUT09/37-26
Record Dates: First submitted 2013-10-11; First posted 2013-11-21 (Estimated); Last update posted 2013-11-21 (Estimated); Status verified 2013-09

CONDITIONS: Hallux Valgus; Pain
Keywords: hallux valgus; pain; functional status; quality of life
MeSH Terms: conditions — Hallux Valgus; Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hallux valgus patients: Females patients with hallux valgus asses for pain, function, and quality of life

SUMMARY:
To investigate relationship between HV deformity and position of rearfoot joints, and its effects on the quality of life, pain, and related functional status in women with bilateral hallux valgus (HV).

DETAILED DESCRIPTION:
To investigate relationship between HV deformity and position of rearfoot joints, and its effects on the quality of life, pain, and related functional status in women with bilateral hallux valgus (HV). Study included 27 right-dominant women. Demographic data, HV angle, weight-bearing and non-weight-bearing subtalar pronation (SP), and navicular height were recorded. Visual Analog Scale, Foot Function Index (FFI), and the American Orthopaedic Foot and Ankle Society (AOFAS) MTP-IP along with AOFAS Mid foot (MF) Scales, and SF-36 were used. HV angle, weight-bearing SP, and pain intensity of the left foot were higher. HV angle of left foot was correlated with all sub-sections of FFI, pain parameter of AOFAS MTP-IP, and pain and total score of AOFAS-MF Scale ). HV angle of left foot was correlated with physical role, pain, and social function sub-domains of SF-36. Right HV angles were correlated with right foot pain and non-weight-bearing SP.Increasing HV angle and pathomechanical changes in rear foot were correlated. Besides, although all participants were right-dominant, their left foot problems were more highlighted.

ELIGIBILITY:
Inclusion Criteria:Inclusion criteria were as follows:

* Women in an age range of 18-55 years,
* Having bilateral deformity with right-dominance,
* First MTP angle of > 15° as radiologically determined by the referring physician,
* Deformity intensity > 2 based on the Manchester scale,
* Muscle forces on ankle and foot > 4
* Having no systemic disease that affects foot biomechanics with no history of surgery,
* Having no neurological problems,
* Having no cognitive, mental, or psychological problems.

Exclusion Criteria:

-

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Effects of hallux valgus deformity in women
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2012-03; Primary Completion 2012-09 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Pain | baseline
  Pain was measured using by Visual Analog Scale
AOFAS Mid foot (MF) Scales | baseline

SECONDARY OUTCOMES:
HV angle and navicular height | baseline
  HV angle was measured by using Universal Goniometers

OTHER OUTCOMES:
Foot Function Index | baseline
  Using the Foot Function Index
American Orthopaedic Foot and Ankle Society (AOFAS)MTP-IP | baseline
weight-bearing and non-weight-bearing subtalar pronation (SP) | baseline
SF-36 | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Burcu TALU, PT. MSc, Study Director — İnönü University, School of Malatya Health, Department of Physiotherapy and Rehabilitation; Gürsoy COŞKUN, PT. PhD., Principal Investigator — Hacettepe University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Ankara, TURKEY; Nilgün BEK, PT. PhD., Study Chair — Hacettepe University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Ankara, TURKEY; Kezban BAYRAMLAR, PT. PhD, Study Chair — Hacettepe University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Ankara, TURKEY

REFERENCES:
- [Background] Coughlin MJ, Jones CP. Hallux valgus: demographics, etiology, and radiographic assessment. Foot Ankle Int. 2007 Jul;28(7):759-77. doi: 10.3113/FAI.2007.0759. PMID 17666168
- [Background] Bock P, Kristen KH, Kroner A, Engel A. Hallux valgus and cartilage degeneration in the first metatarsophalangeal joint. J Bone Joint Surg Br. 2004 Jul;86(5):669-73. doi: 10.1302/0301-620x.86b5.14766. PMID 15274261
- [Background] Robinson AH, Limbers JP. Modern concepts in the treatment of hallux valgus. J Bone Joint Surg Br. 2005 Aug;87(8):1038-45. doi: 10.1302/0301-620X.87B8.16467. No abstract available. PMID 16049235
- [Background] Menz HB, Lord SR. Foot problems, functional impairment, and falls in older people. J Am Podiatr Med Assoc. 1999 Sep;89(9):458-67. doi: 10.7547/87507315-89-9-458. PMID 10507214
- [Background] Coughlin MJ. Hallux valgus. J Bone Joint Surg Am. 1996 Jun;78(6):932-66. No abstract available. PMID 8666613
- [Background] Bek N, Kürklü B. Comparison of the effects of different conservative treatment methods in treatment of hallux valgus. [Halluks valgus tedavisinde kullanılan farklı konservatif yöntemlerin etkinliklerinin karşılaştırılması.] Article in Turkish. Artroplasti Artroskopik Cerrahi 2002;13:90-93.
- [Background] Coughlin MJ. Hallux valgus. Causes, evaluation, and treatment. Postgrad Med. 1984 Apr;75(5):174-8, 183, 186-7. doi: 10.1080/00325481.1984.11698000. No abstract available. PMID 6709527
- [Background] Uchiyama E, Kitaoka HB, Luo ZP, Grande JP, Kura H, An KN. Pathomechanics of hallux valgus: biomechanical and immunohistochemical study. Foot Ankle Int. 2005 Sep;26(9):732-8. doi: 10.1177/107110070502600911. PMID 16174504
- [Background] Coughlin MJ, Thompson FM. The high price of high-fashion footwear. Instr Course Lect. 1995;44:371-7. No abstract available. PMID 7797875
- [Background] Roddy E, Zhang W, Doherty M. Prevalence and associations of hallux valgus in a primary care population. Arthritis Rheum. 2008 Jun 15;59(6):857-62. doi: 10.1002/art.23709. PMID 18512715
- [Background] Mann RA, Coughlin MJ. Hallux valgus--etiology, anatomy, treatment and surgical considerations. Clin Orthop Relat Res. 1981 Jun;(157):31-41. PMID 7249460
- [Background] Dawson J, Thorogood M, Marks SA, Juszczak E, Dodd C, Lavis G, Fitzpatrick R. The prevalence of foot problems in older women: a cause for concern. J Public Health Med. 2002 Jun;24(2):77-84. doi: 10.1093/pubmed/24.2.77. PMID 12141589
- [Background] SIM-FOOK L, HODGSON AR. A comparison of foot forms among the non-shoe and shoe-wearing Chinese population. J Bone Joint Surg Am. 1958 Oct;40-A(5):1058-62. No abstract available. PMID 13587573
- [Background] BARNICOT NA, HARDY RH. The position of the hallux in West Africans. J Anat. 1955 Jul;89(3):355-61. No abstract available. PMID 13251965
- [Background] Menz HB, Morris ME. Footwear characteristics and foot problems in older people. Gerontology. 2005 Sep-Oct;51(5):346-51. doi: 10.1159/000086373. PMID 16110238
- [Background] Piggott H. The natural history of hallux valgus in adolescence and early adult life. J Bone Joint Surg. 1960;42(B):749-60.
- [Background] Saro C, Jensen I, Lindgren U, Fellander-Tsai L. Quality-of-life outcome after hallux valgus surgery. Qual Life Res. 2007 Jun;16(5):731-8. doi: 10.1007/s11136-007-9192-6. Epub 2007 Mar 7. PMID 17342454
- [Background] Abhishek A, Roddy E, Zhang W, Doherty M. Are hallux valgus and big toe pain associated with impaired quality of life? A cross-sectional study. Osteoarthritis Cartilage. 2010 Jul;18(7):923-6. doi: 10.1016/j.joca.2010.03.011. Epub 2010 Apr 22. PMID 20417286
- [Background] Menz HB, Roddy E, Thomas E, Croft PR. Impact of hallux valgus severity on general and foot-specific health-related quality of life. Arthritis Care Res (Hoboken). 2011 Mar;63(3):396-404. doi: 10.1002/acr.20396. Epub 2010 Nov 15. PMID 21080349
- [Background] Lazarides SP, Hildreth A, Prassanna V, Talkhani I. Association amongst angular deformities in halluks valgus and impact of the deformity in health-related quality of life. Foot and Ankle Surgery. 2005;11:193-6.
- [Background] Annett M. The distribution of manual asymmetry. Br J Psychol. 1972 Aug;63(3):343-58. doi: 10.1111/j.2044-8295.1972.tb01282.x. No abstract available. PMID 4199291
- [Background] Karadağ A, Kutlu M. Effects of long-term football exercises on auido-visual reaction times on players' dominant and non-dominant feet [Uzun dönem futbol antrenmanların futbolcuların baskın ve baskın olmayan ayaklarının görsel işitsel reaksiyon zamanlarına etkileri]. Article in Turkish. Fırat Tıp Dergisi. 2006;11:26-29.
- [Background] Gabbard C. Foot laterality during childhood: a review. Int J Neurosci. 1993 Oct;72(3-4):175-82. doi: 10.3109/00207459309024106. PMID 8138373
- [Background] Garrow AP, Papageorgiou A, Silman AJ, Thomas E, Jayson MI, Macfarlane GJ. The grading of hallux valgus. The Manchester Scale. J Am Podiatr Med Assoc. 2001 Feb;91(2):74-8. doi: 10.7547/87507315-91-2-74. PMID 11266481
- [Background] Mendell JR, Florence J. Manual muscle testing. Muscle Nerve. 1990;13 Suppl:S16-20. doi: 10.1002/mus.880131307. No abstract available. PMID 2233877
- [Background] Lamur KS, Huson A, Snijders CJ, Stoeckart R. Geometric data of hallux valgus feet. Foot Ankle Int. 1996 Sep;17(9):548-54. doi: 10.1177/107110079601700907. PMID 8886782
- [Background] Gajdosik RL, Bohannon RW. Clinical measurement of range of motion. Review of goniometry emphasizing reliability and validity. Phys Ther. 1987 Dec;67(12):1867-72. doi: 10.1093/ptj/67.12.1867. PMID 3685114
- [Background] Giladi M, Milgrom C, Stein M. The low arch: A protective factor in stress fractures: A prospective study of 295 military recruits. Orthop Rev. 1985;14:81-4.
- [Background] Dahle LK, Mueller MJ, Delitto A, Diamond JE. Visual assessment of foot type and relationship of foot type to lower extremity injury. J Orthop Sports Phys Ther. 1991;14(2):70-4. doi: 10.2519/jospt.1991.14.2.70. PMID 18796826
- [Background] Hills AP, Hennig EM, McDonald M, Bar-Or O. Plantar pressure differences between obese and non-obese adults: a biomechanical analysis. Int J Obes Relat Metab Disord. 2001 Nov;25(11):1674-9. doi: 10.1038/sj.ijo.0801785. PMID 11753590
- [Background] Knutzen KM, Price A. Lower extremity static and dynamic relationships with rearfoot motion in gait. J Am Podiatr Med Assoc. 1994 Apr;84(4):171-80. doi: 10.7547/87507315-84-4-171. PMID 8201551
- [Background] McPoil T, Cornwall MW. Relationship between neutral subtalar joint position and pattern of rearfoot motion during walking. Foot Ankle Int. 1994 Mar;15(3):141-5. doi: 10.1177/107110079401500309. PMID 7951942
- [Background] Menz HB. Alternative techniques for the clinical assessment of foot pronation. J Am Podiatr Med Assoc. 1998 Mar;88(3):119-29. doi: 10.7547/87507315-88-3-119. PMID 9542353
- [Background] Gallagher EJ, Liebman M, Bijur PE. Prospective validation of clinically important changes in pain severity measured on a visual analog scale. Ann Emerg Med. 2001 Dec;38(6):633-8. doi: 10.1067/mem.2001.118863. PMID 11719741
- [Background] Agel J, Beskin JL, Brage M, Guyton GP, Kadel NJ, Saltzman CL, Sands AK, Sangeorzan BJ, SooHoo NF, Stroud CC, Thordarson DB. Reliability of the Foot Function Index:: A report of the AOFAS Outcomes Committee. Foot Ankle Int. 2005 Nov;26(11):962-7. doi: 10.1177/107110070502601112. PMID 16309612
- [Background] Baumhauer JF, Nawoczenski DA, DiGiovanni BF, Wilding GE. Reliability and validity of the American Orthopaedic Foot and Ankle Society Clinical Rating Scale: a pilot study for the hallux and lesser toes. Foot Ankle Int. 2006 Dec;27(12):1014-9. doi: 10.1177/107110070602701202. PMID 17207425
- [Background] Koçyiğit H, Aydemir Ö, Ölmez N, Memiş A. Turkish reliability and validity of SF-36. [SF-36 nın Türkçe için güvenilirliği ve geçerliliği.] Article in Turkish. İlaç ve Tedavi Dergisi 1999;12:102-6.
- [Background] Budiman-Mak E, Conrad KJ, Roach KE. The Foot Function Index: a measure of foot pain and disability. J Clin Epidemiol. 1991;44(6):561-70. doi: 10.1016/0895-4356(91)90220-4. PMID 2037861
- [Background] SooHoo NF, Shuler M, Fleming LL; American Orthopaedic Foot and Ankle Society. Evaluation of the validity of the AOFAS Clinical Rating Systems by correlation to the SF-36. Foot Ankle Int. 2003 Jan;24(1):50-5. doi: 10.1177/107110070302400108. PMID 12540082
- [Background] Tüzün Ç, Tıkız C. Foot problems in the elderly. Turkish Journal of Geriatrics. 2003;6:135-41.
- [Background] Scott G, Menz HB, Newcombe L. Age-related differences in foot structure and function. Gait Posture. 2007 Jun;26(1):68-75. doi: 10.1016/j.gaitpost.2006.07.009. Epub 2006 Sep 1. PMID 16945538
- [Background] HARDY RH, CLAPHAM JC. Observations on hallux valgus; based on a controlled series. J Bone Joint Surg Br. 1951 Aug;33-B(3):376-91. doi: 10.1302/0301-620X.33B3.376. No abstract available. PMID 14861244
- [Background] Nork SE, Coughlin RR. How to examine a foot and what to do with a bunion. Prim Care. 1996 Jun;23(2):281-97. doi: 10.1016/s0095-4543(05)70276-1. PMID 8784930
- [Background] Wong YS. Influence of the abductor hallucis muscle on the medial arch of the foot: a kinematic and anatomical cadaver study. Foot Ankle Int. 2007 May;28(5):617-20. doi: 10.3113/FAI.2007.0617. PMID 17559771